CLINICAL TRIAL: NCT02484170
Title: Mannitol Cream in the Treatment of Post-herpeticNeuralgia;a Randomized Placebo-Controlled Crossover Pilot Study
Brief Title: Mannitol Cream for Post Herpetic Neuralgia
Acronym: MannitolPHN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Helene Bertrand, MD, CCFP, Clinical instructor, Department of family practice University of British Columbia, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H15-01260
Record Dates: First submitted 2015-06-13; First posted 2015-06-29 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Neuralgia, Postherpetic
Keywords: Mannitol; cream; neuropathic pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — Mannitol

STUDY DESIGN:
Intervention Model Description: 1 week observation, one week cream A assigned, 3 day crossover, one week of cream B assigned. After the crossover study, 3 months of mannitol cream assigned.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mannitol in vehicle cream /vehicle cream (Active Comparator): one week on the mannitol cream (mannitol 30% in vehicle cream), a 3 day washout period, and one week on the placebo cream (vehicle cream alone). To be applied over the painful area as needed for pain. Usual frequency is 2 to 3 times daily.
  Interventions: Drug: Mannitol cream; Drug: Placebo
- vehicle cream /mannitol in vehicle cream (Active Comparator): one week on the placebo cream (vehicle cream alone), a 3 day washout period, and one week on the mannitol cream (mannitol 30% in vehicle cream).To be applied over the painful area as needed for pain. Usual frequency is unknown.
  Interventions: Drug: Mannitol cream; Drug: Placebo

INTERVENTIONS:
Drug: Mannitol cream — Apply to area of postherpetic neuralgia pain as needed for pain control. Usual frequency is 2 to 3 times per day.For crossover study, will be applied for 7 days. For observational study, will be applied up to 3 months
  Other Names: Mannitol in vehicle cream; QR cream
Drug: Placebo — Apply to area of postherpetic neuralgia pain as needed for pain control.Usual frequency is unknown. For crossover study, will be applied for 7 days. Will not be used after crossover study
  Other Names: Vehicle cream

SUMMARY:
30% mannitol cream has shown its ability to reduce the activation of the Capsaicin (TRPV1) (Transient Receptor Potential Vanilloid 1) receptor, a likely cause of the pain of post-herpetic neuralgia (PHN). This randomized placebo-controlled crossover study compares PHN pain one week before, for one week on the randomly assigned mannitol versus placebo cream and, after a three day washout, for one week on the other cream. Following this crossover study, participants receive mannitol cream for three months. Pain levels will be checked to assess whether continued use of this cream significantly reduces the pain levels associated with PHN. If pain persists beyond 3 months, participants will be offered mannitol and menthol cream for one month following which their pain levels will be checked.

DETAILED DESCRIPTION:
Pain levels: 0 to 10 Numerical Rating Scale (NRS), medication and alcohol intake will be checked daily for one week prior to randomization in 20 participants with post herpetic neuralgia, lasting more than three months. Following this 10 will be randomized to apply 30% mannitol in vehicle cream and 10 to apply vehicle cream alone for one week during which daily pain levels and use of medication and alcohol will be measured together with the mode of application (rubbing in or applying it to cling wrap then applying the cream coated cling wrap to the skin in cases of severe allodynia). After a three day washout period, they will be given the cream they did not receive previously for one week. The same variables will be recorded daily. The data collected in the first 24 days will be used to generate a power analysis. Following this, all subjects will receive the 30% mannitol cream to apply for three months. Their pain levels, medication intake and method of application will be measured once a month for three months. T-tests will compare the pain levels for mannitol and placebo users before and after one week of the use of each cream to see if the mannitol cream provides better short term pain relief than placebo. Repeated measures ANOVA (Analysis Of VAriance) will compare pain levels before using the mannitol cream and monthly for three months to assess the long-term effects of mannitol cream. Variables collected at each visit, which will not be used for statistical purposes in the current very small pilot project but may be used in a later study, include: application method, effect and side effects of the cream, medication and alcohol use, PHQ - 9 (Personal Health Questionnaire, 9 questions), and questions from the brief pain inventory score. At three months, a satisfaction score will be added to the database. If pain persists beyond 3 months, participants will be offered mannitol and menthol cream for one month, following which their pain levels, PHQ - 9 and brief pain inventory scores will be checked.

ELIGIBILITY:
Inclusion Criteria

1. - Suffering from post-herpetic neuralgia on the trunk or the extremities for at least three months.
2. - Maximum daily pain score greater than or equal to 5/10.
3. - Having failed to improve with at least one neuropathic pain medication.

4- Able and willing to fill a fluid survey NRS pain scale and a medication intake questionnaire daily, preferably online but on paper, if unable, for the first 24 days of the study, then once a month for three months..

5 - Preferably have access to someone who can apply cream to their back if they have pain in the back and cannot reach the area.

6 - If that is not possible, ability to apply the cream to their own back, using an applicator which will be supplied.

Exclusion Criteria:

1. Allergies to any of the ingredients of the cream
2. Open lesions or abrasions on the skin where the cream will be applied
3. Using corticosteroids
4. Unwilling to stop using other topical products (creams or patches) for the treatment of post-herpetic neuralgia
5. Pregnant, breast-feeding or not using birth control
6. Suffering from severe chronic pain from a cause other than post-herpetic neuralgia

   -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-30; Primary Completion 2016-04-29 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Change in worst NRS (Numerical Rating Scale) pain score | Before each cream is first applied, 7 days later, and for mannitol cream 1,2 and 3 months
  In the last 24 hours, how bad was your pain at its worst? No pain 0 1 2 3 4 5 6 7 8 9 10 Worst pain imaginable
Change in average NRS (Numerical Rating Scale) pain score | Before each cream is first applied, 7 days later, and for mannitol cream 1,2 and 3 months
  In the last 24 hours, how bad was your pain on average? No pain 0 1 2 3 4 5 6 7 8 9 10 Worst pain imaginable

SECONDARY OUTCOMES:
Change in Pain medication intake | Before each cream is first applied, 7 days later, and for mannitol cream 1,2 and 3,months
  Number of pills taken for pain in one day. Will decrease as the pain intensity decreases. Write the number of tablets that you took: 1. Tylenol/acetaminophen______, 2. Anti-inflammatory medication like Advil/ibuprofen, naproxen, diclofenac, Voltaren, Aleve______, 3. Tylenol or ASA (acetylsalicylic acid) plus narcotic like Tylenol 3, or 292 or Tramacet (acetaminophen/tramadol) ______, 4. Narcotic like morphine, hydromorphone/dilaudid, fentanyl, Demerol, tramadol______, 5. Cannabis, marijuana, or pot______, The total in each category will be added to calculate the total number of tablets taken in 24 hours.
Change in Alcohol intake | Before each cream is first applied, 7 days later, and for mannitol cream 1,2 and 3 months
  Number of alcoholic drinks in one day. May decrease as the pain intensity decreases. Write down the total number of alcoholic drinks you had in the last 24 hours:how many glasses of wine ______ glasses of hard liquor______ bottles of beer______. The total number of glasses will be recorded.
Change in questions from the brief pain inventory score | Before each cream is first applied, 7 days later, and for mannitol cream 1,2 and 3 months
  The total from the following questions will be recorded to measure how much their pain is interfering with their lives: Circle one number. In the last 24 hours, how much has your pain interfered with your:
  General activity:, Mood: Walking ability: Normal work: (includes both work outside the home and housework) Relations with other people: Sleep: Enjoyment of life: Each of these will be scored as follows: does not interfere 0 1 2 3 4 5 6 7 8 9 10 completely interferes. The scores added up. This sum should decrease as the pain decreases.
Change in PHQ-9 (Personal health questionnaire, 9 questions) Score | Before each cream is first applied, 7 days later, and for mannitol cream 1,2 and 3 months
  Patients will fill the PHQ - 9 score. http://phqscreeners.com/pdfs/02_PHQ-9/English.pdf The sum of the answers from this questionnaire, which is used to measure the degree of depression, may decrease as the pain intensity decreases.
Change in Method of cream application | when each cream is first applied, 7 days later, and for mannitol cream 1,2 and 3 months
  Patients will describe whether they use cling wrap (4), gentle applicator (3) or rubbing in gently (2) or vigourous rubbing (1)
Change in effect and side effects of the cream | Daily for the 14 days, of the crossover study, then at 1,2 and 3 months
  How many times did you apply the cream today?_______ Circle one number. How bad was your pain?.. Before you applied the cream? NRS 0-10 1hour after you applied the cream? NRS 0-10 Did the cream relieve your pain? No □ if Yes □ in how many minutes?____ For how many hours was your pain relieved?____ Did you experience a side effect from the cream? No □ if Yes □ What was it?_________________ Any comments?_______________________
Satisfaction from cream use | Three months after use of mannitol cream was started.
  How satisfied were you with the use of this cream? Not at all satisfied 0 1 2 3 4 5 6 7 8 9 10 extremely satisfied
Change in pain score from mannitol cream use to mannitol and menthol cream use | 1st measurement Three months after use of mannitol cream was started 2nd measurement one month after mannitol and menthol cream started
  Maximum pain score after 3 months of mannitol cream use compared to maximum pain score after one month of mannitol and menthol cream use

CONTACTS AND LOCATIONS:
Overall Officials: Helene Bertrand, MD, CM, CCFP, Principal Investigator — University of British Columbia, Department of family practice
Locations (1):
- Dr. Helene Bertrand Inc., North Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Bertrand H, Kyriazis M, Reeves KD, Lyftogt J, Rabago D. Topical Mannitol Reduces Capsaicin-Induced Pain: Results of a Pilot-Level, Double-Blind, Randomized Controlled Trial. PM R. 2015 Nov;7(11):1111-1117. doi: 10.1016/j.pmrj.2015.05.002. Epub 2015 May 12. PMID 25978942
- [Background] Gilron I, Baron R, Jensen T. Neuropathic pain: principles of diagnosis and treatment. Mayo Clin Proc. 2015 Apr;90(4):532-45. doi: 10.1016/j.mayocp.2015.01.018. PMID 25841257
- [Background] Shannon HJ, Anderson J, Damle JS. Evidence for interventional procedures as an adjunct therapy in the treatment of shingles pain. Adv Skin Wound Care. 2012 Jun;25(6):276-84; quiz 285-6. doi: 10.1097/01.ASW.0000415345.22307.f3. PMID 22610112
- [Background] Szolcsanyi J, Sandor Z. Multisteric TRPV1 nocisensor: a target for analgesics. Trends Pharmacol Sci. 2012 Dec;33(12):646-55. doi: 10.1016/j.tips.2012.09.002. Epub 2012 Oct 12. PMID 23068431